CLINICAL TRIAL: NCT05731505
Title: The Effect Of Supportive Approach Structured According To Kolcaba Comfort Theory Applied To Parents Of Children With Cerebral Palsy On Child's Comfort, Quality Of Life, And Parent's Self-Efficiency
Brief Title: The Effect Of Supportive Approach According To Kolcaba Comfort Theory Applied To Parents Of Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Bircan Kahraman Berberoglu, research asistant, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Adnan Menderes Universıty
Record Dates: First submitted 2022-12-10; First posted 2023-02-16 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; comfort theory; nursing care
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: experimental, randomized controlled, single-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THE EFFECT OF A SUPPORTIVE APPROACH STRUCTURED ACCORDING TO KOLCABA'S COMFORT THEORY (Experimental): The study group consisted of parents who were given a supportive approach structured according to Kolcaba's Comfort Theory by the researcher.
  Interventions: Behavioral: theory-based education-consulting
- KOLCABA COMFORT THEORY APPLİED TO PARENTS OF CHİLDREN WİTH CEREBRAL PALSY (Experimental): During the training given by the researcher, the children continued their routine education in the rehabilitation center. Although the education to be done is for the child and their parents, the education was given directly to the parents, since the mental perception levels of the children may not be sufficient and mostly children with CP live dependent on their parents. The parent who will be involved in the research is the primary caregiver who is most interested in the child.
  Interventions: Behavioral: theory-based education-consulting

INTERVENTIONS:
Behavioral: theory-based education-consulting — Parents in the study groups were provided with training and support in line with their needs in the educational issues specified in the Family Education-Support Booklet for a Child with Cerebral Palsy. The control group was not trained. Research data were collected using the Child and Parent Information Form, Needs Determination Form, Relaxed Behavior Checklist (KDKL), Quality of Life for Children Parent Form (PIDQ) and Self-Efficacy Scale. The comfort and quality of life of the children in the study group and the self-efficacy of the parents were evaluated before the education, 1 month and 3 months after the education.

SUMMARY:
Purpose: This study was conducted to evaluate the effect of the structured supportive approach given to the parents of children with cerebral palsy according to Kolcaba Comfort Theory on the child's comfort, quality of life and parent's self-efficacy._

H01: According to Kolcaba's Comfort Theory, there is no difference between the comfort scores of the children of parents (study group) to whom the structured supportive approach was applied and the children of the parents who did not apply this approach (control group).

H02: According to Kolcaba's Comfort Theory, there is no difference between the quality of life scores of the children of parents (study group) to whom the structured supportive approach was applied and the children of parents who did not apply this approach (control group).

H03: According to Kolcaba's Comfort Theory, there is no difference between the self-efficacy scores of the parents (study group) who applied the structured supportive approach and the parents who did not apply this approach (control group)_

DETAILED DESCRIPTION:
This is an experimental, randomized controlled, single-blind study. The study was conducted with the parents of children with CP aged 8-16 years, who went to the rehabilitation centers in a randomized controlled manner between 11 October 2021 and 11 November 2022 to receive education and treatment. The sample consisted of 73 parents, the study group (n=35), and the control group (n=38). Parents in the study groups were given education-support in accordance with their needs in the educational topics specified in the Parent Education-Support Booklet for a Child with Cerebral Palsy. The control group was not trained. Research data were collected using the Child and Parent Information Form, the Needs Determination Form, the Comfort Behaviors Checklist (KDKL), the Parent Form of the Quality of Life Scale for Children (PIDQ) and the Self-Efficacy Scale. The comfort and quality of life of the children in the study group and the self-efficacy of the parents were evaluated before, 1 month and 3 months after the education. The control group's data were collected at the same time as the other groups. Descriptive statistics, Pearson chi-square, Fisher exact chi-square, Student-t, and ANOVA were used in the analysis of the data.

ELIGIBILITY:
The criteria for inclusion of children in the study are:

* Having been diagnosed with cerebral palsy,
* Being between the ages of 8-16,
* Being at the level of 1/2/3/4/5 according to the Gross Motor Function Classification System (KMFSS)

The criteria for inclusion of parents in the study are:

* Being at least literate,
* Being able to speak and understand Turkish,
* Having a smart phone and/or internet connection.

The criteria for exclusion of children from the study are:

• Having drug-resistant epilepsy.

The criteria for exclusion of parents from the study are:

* Caring for other dependent people (elderly, disabled, etc.),
* Being pregnant,
* Having a chronic physical illness (heart disease, diabetes mellitus, hypertension, etc.)
* Having a mental illness (major depression, psychosis, etc.),
* Being hearing, seeing or speaking impaired,
* Having a mental disability.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Comfort Behaviors Checklist | on completion of the study, an average of 3 months
  This form is used to evaluate the comfort of patients who are unable to fill out a questionnaire or who have cognitive limitations. It consists of 30 items. High scores indicate a high level of comfort. If all questions are answered, the lowest score that can be obtained from the scale is 25, and the highest score is 100.High scores indicate increased comfort and low scores indicate decreased comfort.
Quality of Life Scale for Children Parent Form | on completion of the study, an average of 3 months
  The scale is a self-report scale and questions the status of children and adolescents regarding quality of life in the last month. The scale consists of four subsections, 23 items in total, in which physical, emotional, social and school-related functionality are questioned. The scale has a five-choice Likert-type response scale (0=never, 1=rarely, 2=sometimes, 3=often, 4=always). The scores obtained from the items are translated linearly as 0=100, 1=75, 2=50, 3=25, 4=0. If all questions are answered, the lowest score that can be obtained from the scale is 25, and the highest score is 100.High scores indicate an increase in quality of life, and low scores indicate a decrease.
Self-Efficiency Scale | on completion of the study, an average of 3 months
  There are 19 items, seven of which are fillers, and are of a five-point Likert type. Respondents were presented with response categories ranging from "strongly disagree" to "strongly agree". In scoring the items, "strongly disagree" gets 1 point and "strongly agree" gets 5 points; High scores indicate high self-efficacy. If all questions are answered, the lowest score that can be obtained from the scale is 19, and the highest score is 95. High scores indicate an increase in self-efficiency, and low scores indicate a decrease.

CONTACTS AND LOCATIONS:
Overall Officials: Hüsniye Çalışır, Prof. Dr., Study Director — Aydın Adnan Menderes Univercity
Locations (1):
- Adnan Menderes Univercity, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No